CLINICAL TRIAL: NCT00615407
Title: A Pilot Evaluation of the Impact of Alcohol Use on Airway Inflammation and Mechanics in Asthmatics
Acronym: AIM Asthma
Status: Withdrawn | Type: Observational
Why Stopped: Dr. Holguin is relocating.
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00001136
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Asthma
Keywords: Asthma, alcohol
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine, and exhaled breath condensate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alcohol Drinkers: Asthmatics who consume 3 or more alcoholic beverages per day (on average)
- Non Drinkers: Asthmatics who do not drink alcohol or consume less than or equal to 2 alcoholic beverages per month

SUMMARY:
Since 1980, the number of people in the United States diagnosed with asthma has increased dramatically. Studying what causes and triggers asthma is an important part of understanding and subsequently managing this disease. Although some have suggested that alcohol consumption may affect asthma, little is known about how consistent alcohol use affects the amount of inflammation present in the lungs and whether consistent alcohol use makes the airways more narrow and stiff.

Participation in this study involves 2 visits in order to complete questionnaires, various pulmonary function tests, as well as the collection of blood, urine, and exhaled breath condensate specimens.

This study includes optional genetic and bronchoscopy substudies.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Literate in English (i.e., read study materials at 6th grade level) so as to understand, and complete the ratings scales and questionnaires accurately
* Physician-diagnosed asthma requiring treatment in the past year with a post bronchodilator FEV1/FVC >0.70 and at least 12% reversibility after bronchodilator usage
* Alcohol usage groups: 1) those who rarely or who do not drink alcohol (≤2 drinks per month); or 2) those who drink 3 or more alcoholic beverages per day on average

Exclusion Criteria:

* Social drinkers (>2 drinks in a month but <3 drinks per day)
* Asthma exacerbation within the past month
* Current upper respiratory infection
* Active allergies with uncontrolled symptoms
* Current DSM-IV diagnosis of illicit substance dependence (not alcohol)
* History of serious pulmonary problems other than asthma
* Other significant non-pulmonary comorbidities
* Pregnancy or currently lactating
* Daily use of Prednisone or other corticosteroids
* Tobacco smoking within the past year or >10 life-time pack-years of smoking
* Positive breath alcohol level at the time of the study assessments
* Positive urine cotinine test at enrollment (indicates nicotine usage)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, 40 non-smoking adults with asthma will be recruited-50% will be non-drinking and 50% will be heavy alcohol users (≥3 standard drinks/day on average).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Measurements of airway oxidative stress (increased GSSG/GS, and RNS/NO ratios and higher exhaled 8-isoprostanes levels) | single timepoint

SECONDARY OUTCOMES:
Measurements of lung function (spirometry, response to methacholine challenge, and impulse oscillometry). | single timepoint
Asthma symptoms and control through standard asthma questionnaires | single timepoint